CLINICAL TRIAL: NCT01525537
Title: Comparison of Surgical Pleth Index Guided Analgesia With Standard Clinical Practise During Balanced Anesthesia
Brief Title: Surgical Pleth Index (SPI) Guided Analgesia During Sevoflurane Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Berthold Bein, Prof. Dr. med., University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPI-134-2
Record Dates: First submitted 2012-01-26; First posted 2012-02-03 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Balanced Anesthesia
Keywords: Anesthesia General; Anesthetics Inhalation; Diagnostic techniques and procedures
MeSH Terms: interventions — Sufentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPI guided arm (Experimental): sufentanil was adjusted to SPI level
  Interventions: Drug: administration of sufentanil
- Standard practise (Active Comparator): Sufentanil was given at standard practise
  Interventions: Drug: sufentanil

INTERVENTIONS:
Drug: administration of sufentanil — 10 microgram sufentanil were given when SPI above 50 for more then 20 sec
  Arms: SPI guided arm
Drug: sufentanil — sufentanil was given at standard practise
  Arms: Standard practise

SUMMARY:
The aim of the present study was to compare SPI guided analgesia with standard clinical practise during general anesthesia using a balanced setting of sevoflurane and sufentanil anesthesia. It was to be tested whether SPI guided analgesia leads to more cardiovascular stability, less use of analgetics and shorter recovery from anesthesia.

DETAILED DESCRIPTION:
General anesthesia can be considered as a combination of hypnosis, antinociception, and immobility. The monitoring of hypnosis and immobility has been established in clinical practise, however for the evaluation of antinociception a valid monitoring is missing.

The Surgical Pleth Index (SPI; former named Surgical Stress Index-SSI) is a multivariate index derived non invasively from finger plethysmographic signal. It has been demonstrated to correlate with surgical stress intensity. In the setting of total intravenous anesthesia TIVA our group could show beneficial effects of SPI guided analgesia in terms of remifentanil consumption, hemodynamic stability and incidence of unwanted events.

Therefore, we wanted examine whether these beneficial effects of SPI guided anesthesia can be transferred to a setting of balanced anesthesia using a volatile anesthetic sevoflurane and the opioid sufentanil.

The following hypotheses have been made:

1. SPI guided analgesia will result in less sufentanil consumption
2. SPI guided analgesia will result in more hemodynamic stability and faster recovery of the patient after anesthesia, and less opioid use in post operative period

ELIGIBILITY:
Inclusion Criteria:

* age between 18 - 65 years
* ASA physical status I or II
* elective surgery under general anesthesia of 1-2 hours
* written informed consent

Exclusion Criteria:

* pregnancy
* history of cardiac arrhythmia
* presence of any neuromuscular opr neurologic disease
* use of CNS active medication or alcohol/illicit drug abuse -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Sufentanil consumption | during induction and end of anesthesia (1-3 hours)
  We will measure the sufentanil consumption during beginning of anesthesia and extubation in microgram per hour.

SECONDARY OUTCOMES:
hemodynamic stability | from beginning of anesthesia until discharge to ward (1day)
  Hemodynamic stability is measured as number of the following events during anesthesia: hypotension, hypertension, tachykardia, bradykardia.

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Bein, MD, PhD, Study Chair — University Hospital Schleswig-Holstein; Matthias Gruenewald, MD, Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- University Hospital Kiel, Dept. of Anesthesiology and Intensive Care Med., Kiel, Germany

REFERENCES:
- [Background] Chen X, Thee C, Gruenewald M, Wnent J, Illies C, Hoecker J, Hanss R, Steinfath M, Bein B. Comparison of surgical stress index-guided analgesia with standard clinical practice during routine general anesthesia: a pilot study. Anesthesiology. 2010 May;112(5):1175-83. doi: 10.1097/ALN.0b013e3181d3d641. PMID 20418698
- [Background] Gruenewald M, Meybohm P, Ilies C, Hocker J, Hanss R, Scholz J, Bein B. Influence of different remifentanil concentrations on the performance of the surgical stress index to detect a standardized painful stimulus during sevoflurane anaesthesia. Br J Anaesth. 2009 Oct;103(4):586-93. doi: 10.1093/bja/aep206. Epub 2009 Jul 31. PMID 19648155
- [Derived] Gruenewald M, Willms S, Broch O, Kott M, Steinfath M, Bein B. Sufentanil administration guided by surgical pleth index vs standard practice during sevoflurane anaesthesia: a randomized controlled pilot study. Br J Anaesth. 2014 May;112(5):898-905. doi: 10.1093/bja/aet485. Epub 2014 Feb 16. PMID 24535604